CLINICAL TRIAL: NCT05917015
Title: A Clinical Study to Determine if Beta-glucan Reduces the Incidence, Duration or Severity of Upper Respiratory Tract Infections Among Skiers
Brief Title: A Clinical Study to Determine if Beta Glucan Reduces the Incidence, Duration or Severity of URTIs Among Skiers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: USANA Health Sciences (Industry)
Responsible Party: Principal Investigator, Mark Levy, Principal Investigator, USANA Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202206CT
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Upper Respiratory Tract Infections; Mental Stress
MeSH Terms: conditions — Respiratory Tract Infections; Stress, Psychological | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Treatment (Placebo Comparator): a placebo tablet (microcrystalline cellulose) identical in size, shape and color to the treatment
  Interventions: Other: Placebo
- Dietary supplement intervention (Experimental): Participants were treated with 2 beta-glucan containing tablets per day for a total duration of 6 weeks.
  Interventions: Dietary Supplement: Treatment

INTERVENTIONS:
Dietary Supplement: Treatment — Participants will receive daily 2 tablets of Proglucamune for a duration of 6 weeks. Each tablet contains ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
  Other Names: Treatment brand name: Proglucamune (USANA Health Sciences)
  Arms: Dietary supplement intervention
Other: Placebo — Participants will receive daily 2 placebo tablets containing microcrystalline cellulose. The size, shape and appearance of the placebo tablet is identical to the treatment tablet.
  Arms: Placebo Treatment

SUMMARY:
This study is designed to determine if a dieatary supplement containing beta-glucan can reduce the incidence, severity and duration of upper respiratory tract infections among a group of highly trained athletes

DETAILED DESCRIPTION:
In this study, we hypothesize that consumption of 200 mg beta-glucan per day will lessen the frequency, duration and severity of URTI symptoms in a population of elite, internationally competitive skiers over a 45-day period. In order to complete this objective, we will utilize the Wisconsin Upper Respiratory Symptom Survey-24 (WURSS-24) to monitor and quantify the incidence, duration and severity of URTI symptoms. A secondary objective is to determine if beta-glucan supplementation reduces or mitigates early indictors of athlete-specific stress. This objective will be assessed using the Athlete Psychological Strain Questionnaire (APSQ), a 10-question patient-reported outcome tool used to evaluate athlete-specific psychological stress.

This will be a randomized, double blind, placebo controlled, parallel arm design conducted over a 6-week period. 50-60 healthy subjects will be recruited and randomized in a 1:1 ratio to either of two interventions:

1. Placebo: daily consumption of the placebo tablet
2. Treatment: daily consumption of the supplement (treatment) tablet

In addition, subjects will complete the WURSS-24 survey daily, and the APSQ survey weekly.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent by signing the electronic Information and Consent Form.
* Male or females between the ages of 18 and 30 (inclusive) without regard to race or ethnic background
* Are in generally good health and have no medical conditions that would prevent or interfere with their participation in the study
* Are fully able and willing to comply with the requirements of the study
* Are fully able and willing to keep scheduled appointments

Exclusion Criteria:

* Females that are pregnant, attempting to become pregnant or are currently lactating/nursing a child.
* Individuals currently taking prescription medications that are known to be immunosuppressants (e.g. dexamethasone, tacrolimus, methotrexate)
* Individuals with gastrointestinal conditions (e.g., inflammatory bowel disease, Crohn's disease, etc.) that may affect consumption of the treatment supplements.
* Individuals with clinically important renal, hepatic, cardiac pulmonary, pancreatic, neurologic or biliary disorders; insulin-dependent and orally controlled diabetics will also be excluded from the study.
* Individuals with a recent history of cancer other than non-melanoma skin cancer.
* Individual's that have trouble swallowing pills.
* Individuals that have participated as a subject in any other clinical study within 30 days of screening.
* Individuals with a history of alcohol abuse or other substance abuse within the previous 2 years.
* Individuals that currently use tobacco products including chewing tobacco and cigarettes.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper respiratory tract symptoms | 6 weeks
  The frequency, duration and severity of upper respiratory tract symptoms among study participants will be monitored via a self reported questionnaire administered daily.

SECONDARY OUTCOMES:
Athlete psychological stress | 6 weeks
  The degree of athlete psychological stress symptoms among study participants will be monitored via a self reported questionnaire administered weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levy, PhD, Principal Investigator — USANA Health Sciences
Locations (1):
- US Ski and Snowboard Center of Excellence, Park City, Utah, United States